CLINICAL TRIAL: NCT05235646
Title: Detection of the Occurrence of Infiltration of Gadolinium Injection in Brain MR Scans Using Artificial Intelligence
Brief Title: Infiltration of Gadolinium Injection in Brain MR Scans Using Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James G. Pipe, Principal Investigator, Mayo Clinic
Other Study IDs: 21-010301
Record Dates: First submitted 2022-01-19; First posted 2022-02-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to develop machine learning algorithms to analyze images from brain MRI to confirm that contrast agent has been correctly administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a MR brain without and with contrast examination on any GE or Siemens 1.5T and 3T MRI system within Mayo Clinic, Rochester, as part of their care plan.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing MR brain without and with IV contrast examination as part of their care plan.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Detection of Infiltration of Gadolinium contrast agent into tissue and muscle using artificial intelligence model | 2 months
  Correct detection of the presence of infiltration of Gadolinium contrast agent into tissue and muscleusing an artificial intelligence model. This outcome will be determined by measuring the difference in signal enhancement in the nasal mucosa or the lack of signal enhancement within the nasal mucosa.

CONTACTS AND LOCATIONS:
Overall Officials: James Pipe, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Study Protocol (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT05235646/Prot_000.pdf